CLINICAL TRIAL: NCT02031536
Title: A Randomized, Double-Blinded, Placebo-Controlled Phase II Study of Adjuvant Everolimus Following the Resection of Metastatic Pancreatic Neuroendocrine Tumors to the Liver
Brief Title: Everolimus in Patients With Pancreatic Neuroendocrine Tumors Metastatic to the Liver Previously Treated With Surgery
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: E2212; NCI-2013-02484 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); ECOG-E2212 (Other: ECOG-ACRIN); U10CA021115 (NIH)
Record Dates: First submitted 2014-01-07; First posted 2014-01-09 (Estimated); Results first posted 2020-12-02 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Gastrinoma; Glucagonoma; Insulinoma; Liver Metastases; Pancreatic Polypeptide Tumor; Recurrent Islet Cell Carcinoma; Somatostatinoma
Keywords: everolimus; randomized; metastatic pancreatic neuroendocrine tumors; liver
MeSH Terms: conditions — Gastrinoma; Glucagonoma; Insulinoma; Carcinoma, Islet Cell; Somatostatinoma | interventions — Everolimus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No

ARMS (2):
- Arm A (everolimus) (Experimental): Patients receive everolimus PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: everolimus
- Arm B (placebo) (Placebo Comparator): Patients receive placebo PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: placebo

INTERVENTIONS:
Drug: everolimus — Given PO
  Other Names: 42-O-(2-hydroxy)ethyl rapamycin; Afinitor; RAD001
  Arms: Arm A (everolimus)
Other: placebo — Given PO
  Other Names: PLCB
  Arms: Arm B (placebo)

SUMMARY:
This randomized phase II trial studies how well everolimus works in treating patients with pancreatic neuroendocrine tumors metastatic to the liver previously treated with surgery. Everolimus may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Giving everolimus after surgery may kill any tumors cells that remain.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate if the addition of adjuvant everolimus to the R0 or R1 surgical resection of pancreatic neuroendocrine tumor metastases to the liver will result in an improvement in disease free survival.

SECONDARY OBJECTIVES:

I. To evaluate if the addition of adjuvant everolimus to the R0 or R1 surgical resection of pancreatic neuroendocrine tumor metastases to the liver will result in an improvement in overall survival.

II. To evaluate the toxicity associated with adjuvant everolimus following resection in patients with metastatic pancreatic neuroendocrine tumors to the liver.

OUTLINE: Patients are randomized to 1 of 2 treatment arms in a 1:1 ratio.

ARM A: Patients receive everolimus orally (PO) once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

ARM B: Patients receive placebo PO QD on days 1-28. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

PROJECTED ACCRUAL: 150 patients

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients must have histologically or pathologically confirmed metastatic low or intermediate grade pancreatic neuroendocrine tumor(s) to the liver as per the Klimstra guidelines
* Patients must have recovered from an R0 or R1 resection of all disease (including resection of a primary primitive neuroectodermal tumor [PNET] if present); patients may have had resection plus microwave or radiofrequency ablation, provided that no ablated lesion was >= 5 cm prior to ablation
* Patients must be within 4 to 8 weeks from the completion of surgery at time of randomization
* Patients must have paraffin-embedded fixed metastatic tumor tissue available for submission for central review; core biopsy or surgical specimens required
* Patients must have post-operative computed tomography (CT) or magnetic resonance imaging (MRI) prior to randomization and =< 4 weeks after completion of surgery to confirm disease status; patients must be able to tolerate CT or MRI imaging including contrast agents as required for the protocol
* Women of child-bearing potential and sexually active males must be strongly advised to use an accepted and highly effective method of contraception or abstain from sexual intercourse for the duration of their treatment through 8 weeks after their last dose of protocol therapy; women of child-bearing potential, sexually active males, and the female partners of male participants should be advised of the risk of becoming pregnant or fathering a child while receiving protocol treatment; should a woman become pregnant while participating in this study, she should inform her treating physician immediately; if a man impregnates a woman while participating in this study, he should inform his treating physician immediately
* Prior treatment with sunitinib and/or cytotoxic chemotherapy are allowed provided last dose was > 30 days prior to randomization
* Prior chemoembolization is allowed provided last dose was > 30 days prior to randomization
* Total bilirubin =< 1.5 X institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 5 X institutional ULN
* Serum creatinine =< 1.5 X institutional ULN or creatinine clearance >= 60 mL/min for patients with creatinine levels above 1.5 X institutional normal
* Fasting serum cholesterol =< 300 mg/dL OR =< 7.75 mmol/L AND fasting triglycerides =< 2.5 x ULN
* Absolute neutrophil count >= 1,500/mm^3
* Leukocytes >= 3,000/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dL
* Patients with a history of the following within =< 12 months of randomization are not eligible

  * Arterial thromboembolic events
  * Unstable angina
  * Myocardial infarction
* Patients with known history of abnormal pulmonary function must have documentation of diffusing capacity of the lung for carbon monoxide (DLCO) of > 50% predicted and oxygen saturation (SaO2) of > 87% at rest on room air =< 4 weeks prior to randomization
* Patients with unexplained pulmonary infiltrates must have pulmonary function tests within the institutional limits of normal =< 4 weeks prior to randomization
* Patients with poorly controlled diabetes mellitus as defined by hemoglobin A1c (HbA1c) > 8% despite adequate therapy are ineligible; patients with a known history of impaired fasting glucose or diabetes mellitus must have blood glucose and antidiabetic treatment monitored closely throughout the trial and adjusted as necessary
* Patients may not be receiving any other investigational agents while on study treatment; prior treatment with other investigational agent is allowed provided last dose was >= 30 days prior to randomization
* Patients must NOT have received live attenuated vaccines =< 1 week prior to randomization; patients should also be advised not to receive live attenuated vaccines during the study and to avoid close contact with others who have received live attenuated vaccines; examples of live attenuated vaccines include intranasal influenza, measles, mumps, rubella, oral polio, Bacillus Calmette-Guerin (BCG), yellow fever, varicella and TY21a typhoid vaccines
* Patients must have Eastern Cooperative Oncology Group (ECOG) performance status =< 1
* Patients must have life expectancy >= 12 weeks
* Patients should be advised to avoid drugs or foods that are known potent cytochrome P450, family 3, subfamily A, polypeptide 4 (CYP3A4) inhibitors or inducers

EXCLUSION CRITERIA:

* Patients have received prior everolimus
* Patients have either clinically apparent central nervous system metastases or carcinomatous meningitis =< 6 months prior to randomization
* Women are pregnant or breast-feeding; all females of childbearing potential must have a blood test within 2 weeks prior to randomization to rule out pregnancy
* Patients are on chronic treatment with corticosteroids or other immunosuppressive agents; topical or inhaled corticosteroids are allowed
* Patients have history of allergic reactions attributed to compounds of similar chemical or biologic composition to everolimus
* Patients have known intolerance or hypersensitivity to everolimus or other rapamycin analogs (e.g. sirolimus, temsirolimus)
* Patients have absorption issues that would limit the ability to absorb everolimus
* Patients have a history of non-compliance to medical regimens or who are considered potentially unreliable or will not be able to complete the entire study
* Patients have previous or concurrent malignancy; exceptions are made for patients who meet any of the following conditions:

  * Non-melanoma skin cancer, in situ cervical cancer, breast cancer in situ, or superficial bladder cancer (noninvasive papillary carcinoma or carcinoma in situ); OR
  * Prior malignancy completely excised or removed and patient has been continuously disease free for > 5 years
* Patients have severe and/or uncontrolled medical conditions such as:

  * Unstable angina pectoris, symptomatic congestive heart failure, myocardial infarction =< 6 months prior to randomization, serious uncontrolled cardiac arrhythmia, or any other clinically significant cardiac disease
  * Symptomatic congestive heart failure of New York Heart Association class III or IV
  * Active (acute or chronic) or uncontrolled severe infection, liver disease such as cirrhosis, decompensated liver disease, and chronic hepatitis (i.e. quantifiable hepatitis B virus [HBV]-deoxyribonucleic acid [DNA] and/or positive hepatitis B surface antigen [HbsAg], quantifiable hepatitis C virus [HCV]-ribonucleic acid [RNA])
  * Active, bleeding diathesis
* Patients have known history of human immunodeficiency virus (HIV) seropositivity
* Patients have experienced thrombotic events (deep vein thrombosis, pulmonary embolism) =< 3 months prior to randomization
* Patients have liver disease such as cirrhosis, chronic active hepatitis, or chronic persistent hepatitis at randomization; patients at increased risk for hepatitis B or hepatitis C must be screened for hepatitis prior to randomization
* Patients have ongoing cardiac dysrhythmia of National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (v4.0) grade >= 2, uncontrolled atrial fibrillation of any grade, or corrected QT (QTc) interval > 470 msec
* Patients have history of severely impaired pulmonary function for their age

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2014-04-10 (Actual); Primary Completion 2017-07-19 (Actual); Study Completion 2017-07-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven Libutti, Principal Investigator — Eastern Cooperative Oncology Group
Locations (1):
- Ecog-Acrin, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was activated on January 17, 2014, accrued its first patient on April 10, 2014, and closed to accrual on March 30, 2015. Two patients, both from Stanford University, were randomized to the trial.
Period: Overall Study
Arm/Group | Arm A (Everolimus) | Arm B (Placebo)
Started | 2 | 0
Completed | 1 | 0
Not Completed | 1 | 0
Not completed — ineligible | 1 | 0

BASELINE CHARACTERISTICS:
Population: All enrolled patients
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Everolimus) | Arm B (Placebo) | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Customized [Count of Participants; unit: Participants]
  Age between 45-49 | 2 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival (DFS)
Description: DFS is defined as time from randomization to disease recurrence or death, whichever occurred first. Patients who are still alive are censored at the last date of known free of recurrence.
Time Frame: assessed every 12 weeks while on treatment and then every 3 months if < 2 years from study entry; every 6 months up to 5 years from study entry or recurrence, whichever occurred first
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm A (Everolimus) | Arm B (Placebo)
Number analyzed (Participants) | 2 | 0
years | 1.3 [NA to NA] — There are only 2 patients on this study, and the confidence interval for the median can not be calculated. Full range would reveal patient individual data. |

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as time from randomization to death from any cause. Patients who are still alive are censored at the last date of known alive.
Time Frame: assessed every 3 months if < 2 years from study entry, and every 6 months up to 5 years from study entry or death, whichever occurred first
Population: All enrolled patients
Measure: Median (95% Confidence Interval); unit: years
Arm/Group | Arm A (Everolimus) | Arm B (Placebo)
Number analyzed (Participants) | 2 | 0
years | 2.05 [NA to NA] — There are only 2 patients on this study, and the confidence interval for the median can not be calculated.Full range would reveal patient individual data. |

ADVERSE EVENTS:
Time Frame: Adverse events were assessed at the end of each cycle (1 cycle=4 weeks) and at 30 days after the completion of protocol therapy
Description: Only grades 4-5 hematologic events and grades 3-5 non-hematologic events were reportable on this study.
Arm/Group | Arm A (Everolimus) | Arm B (Placebo)
All-Cause Mortality (participants affected / at risk) | 1/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Everolimus) (N=2) | Arm B (Placebo) (N=0)
Aspartate aminotransferase increase (Investigations) | 1 | 0
Neutrophil count decrease (Investigations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol: Study protocol (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02031536/Prot_000.pdf
  • Study Protocol and Statistical Analysis Plan: 9. Statistical Considerations (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02031536/Prot_SAP_002.pdf
  • Informed Consent Form (2014-04-21): https://cdn.clinicaltrials.gov/large-docs/36/NCT02031536/ICF_001.pdf